CLINICAL TRIAL: NCT01114035
Title: Characterization Phenotypic and Genetic Study of the Intestinal Epithelial Dysplasia or TE
Brief Title: Characterization Phenotypic and Genetic Study of the Intestinal Epithelial Dysplasia or Tufting Enteropathy (TE)
Acronym: DEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P 070163; ID RCB 2009-A01522-53 (Other: AFSSAPS)
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Intestinal Epithelial Dysplasia; Tufting Enteropathy
Keywords: intestinal epithelial dysplasia; characterization phenotypic; genetic study; or " tufting enteropathy "
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): intestinal epithelial dysplasia
  Interventions: Genetic: blood samples and skin biopsies
- Control (Other): Children without intestinal epithelial dysplasia
  Interventions: Genetic: Skin biopsies

INTERVENTIONS:
Genetic: blood samples and skin biopsies — to detect mutations
  Arms: Patients
Genetic: Skin biopsies — to detect mutations
  Other Names: to detect mutations
  Arms: Control

SUMMARY:
This PHRC is centred on the intestinal epithelial dysplasia ( DEI) or " tufting enteropathy " or TE the clinical and histo-pathological descriptions of which are specified well to the digestive plan(shot).

DETAILED DESCRIPTION:
The objectives of this PHRC are:

* the phenotypic analysis of the intestinal epithelial dysplasia by clinical and histo-pathological investigations.
* the identification of proteins involved at the intestinal level in the differentiation, the proliferation and the membership of the epithelial cells
* from the phenotypic study, a genetic analysis of type maps by homozygote on the whole genome partner in an approach guided by possible candidate genes
* the study of the genes, chosen according to their location, to their profile of expression, and to their function in touch with the pathogenic hypotheses

ELIGIBILITY:
Inclusion criteria :

Patient sent in the service of Gastroenterology Pediatric Hepatology of the Hospital Necker Enfants Malades for an intestinal transplantation, from 0 to 15 years old presenting:

* A known epithelial dysplasia (Diagnosis established on the clinical and histo-morphological criteria from one or several intestinal biopsies, with or without diagnosis known or suspected in the family). The objectives are the phenotypic characterization of the case and the revealing of markers characteristic immuno-histochemistry which can be of use to the diagnosis and direct to candidate genes
* Or a suspicion of dysplasia epithelial (compatible clinical History(Story) with or without extra-digestive demonstrations(appearances) of type keratinate punctuated superficial (KPS), abnormalities cutanea or atresia CHOANS with atypical digestive histology and without diagnosis known in the family). The objectives are the diagnosis on the basis of the immuno-histochemistry expression and the existence of an infringement(achievement) conjunctival and the phenotypic characterization of the case
* The lit(enlightened) and written consent of both holders of the parental authority must be beforehand obtained as well as that of the patient if it is in age to understand(include).

Exclusion criteria :

* Not membership in a national insurance scheme (beneficiary or legal successor)
* Family not understanding(including) French
* Refusal of one of both relatives(parents)

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
gene identification | 6 months
  identification of different family of genes involved in intestinal dysplasia

SECONDARY OUTCOMES:
mutation identification | 6 months
  Identification of different mutations involved in intestinal dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Goulet, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Necker Hospital, Paris, France